CLINICAL TRIAL: NCT04317924
Title: Use of Polyglycolic Acid Felt for Air-leak Prevention After Lung Resection
Brief Title: Pneumostasis With Use of Bio-absorbable Mesh and Fibrin Sealant in Lung Resection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not available to conduct the research.
Sponsor: Boston Medical Center (Other)
Collaborators: Gunze Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-37652
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Air Leak From Lung
Keywords: Pneumostasis; Bio-absorbable mesh; Lung resection; Neoveil
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Stratified block randomization will be done using known predictors of prolonged air leak: 1) surgical procedure (wedge vs lobectomy) and 2) presence of pulmonary comorbidities (chronic obstructive pulmonary disease and emphysema).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reinforcement of air leak (Experimental): Participants in this arm will receive reinforcement with the NEOVEIL (polyglycolic acid felt) which will be impregnated with human fibrinogen and thrombin.
  Interventions: Device: Polyglycolic acid felt
- No reinforcement of air leak (Active Comparator): Participants in this arm will receive standard of care for air leak post lung resection.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Polyglycolic acid felt — Neoveil is a polyglycolic acid felt that has been shown to decrease the incidence of prolonged air leak after lung resection in Japan.
  Other Names: Neoveil
  Arms: Reinforcement of air leak
Other: Standard of care — Standard of care after air leak post lung resection
  Arms: No reinforcement of air leak

SUMMARY:
Prolonged air leak, defined as air leak present 5 days after lung resection, is one of the most common complications after lung resection. This leads to patient discomfort (as the chest tube has to stay in place while air leak is present), prolonged stay, and increased cost.

NeoVeil is a bioabsorbable glycolic acid which has been used in Japan and other Asian countries for air leak prevention after lung resections. NeoVeil is impregnated with fibrin sealant materials and is placed on the lung surface at the time of operation. It then acts as a scaffold on resected area which is prone to air leak.

This randomized clinical trial will be the first in the United States to test its efficacy for air leak prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective lung resection at BMC
* Intra-operative diagnosis of air leak

Exclusion Criteria:

* Patients undergoing emergency lung resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Time to removal of chest tubes | 2 years
  The time in hours to removal of chest tubes post lung resection will be abstracted from the electronic medical record of each participant.

SECONDARY OUTCOMES:
Length of hospital stay | 2 years
  The length of hospital stay in days will be abstracted from the electronic medical record of each participant.
Number of participants with additional interventions for air leak | 2 years
  The number of participants requiring additional interventions post lung resection will be abstracted from the electronic medical record of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Kei Suzuki, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No